CLINICAL TRIAL: NCT01587456
Title: Relationship Between Osteoporosis and Arterial Rigidity Within Fractured Patients Cohort.
Brief Title: Arteos II Study: Relationship Between Osteoporosis and Arterial Rigidity Within Fractured Patients Cohort
Acronym: ARTEOS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00453-38
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Osteoporosis
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators planned to study relationship between osteoporosis and arterial rigidity within fractured patients cohort.

ELIGIBILITY:
Inclusion Criteria:

* women and men > 60 years of age
* medical history of low energy fracture
* DXA Tscore -2,5 DS
* FREE AND INFORMED CONSENT SIGNED

Exclusion Criteria:

* women and men < 60 years of age
* Corticoids treatment
* Breast cancer or prostat cancer medical history
* High energy fracture (traumatic fracture)
* No social security affiliation
* Incapacity to informed consent signed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men > 60 years of age with medical history of low energy fracture andradiologic osteoporosis with DXA Tscore at -2,5 DS.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Georges WERYHA, Professor, Principal Investigator — CHU de Brabois Endocrinology
Locations (1):
- CHU de Brabois Endocrinology, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided